CLINICAL TRIAL: NCT05768776
Title: To Compare the Effectiveness of the MOSES 2.0 Technology to the Non-MOSES Technology on the Success Rate of Holmium LASER Enucleation of the Prostate (HoLEP) Performed on an Outpatient Basis in the Context of Benign Prostatic Hypertrophy.
Brief Title: Outpatient Holmium LASER Enucleation of the Prostate: Benefit of MOSES(TM) 2.0 Technology
Acronym: MOSES
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2022/48
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hypertrophy; Holmium Laser Enucleation of the Prostate
Keywords: Benign Prostatic Hypertrophy; HoLEP; MOSES(TM) 2.0; Ambulatory; Men
MeSH Terms: conditions — Prostatic Hyperplasia; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HoLEP patients without MOSESTM 2.0 effect (open label): control retrospective open label
  Interventions: Procedure: HoLEP patients without MOSES(TM) 2.0 effect (open label)
- HoLEP patients with MOSESTM 2.0 effect (open label): prospective open label
  Interventions: Procedure: HoLEP patients with MOSES(TM) 2.0 effect (open label)

INTERVENTIONS:
Procedure: HoLEP patients without MOSES(TM) 2.0 effect (open label) — HoLEP surgery for the treatment of Benign Prostate Hyperthrophy, without using MOSES technology
  Groups: HoLEP patients without MOSESTM 2.0 effect (open label)
Procedure: HoLEP patients with MOSES(TM) 2.0 effect (open label) — HoLEP surgery for the treatment of Benign Prostate Hyperthrophy, with the use of MOSES technology
  Groups: HoLEP patients with MOSESTM 2.0 effect (open label)

SUMMARY:
The aim of this study is to compare the success rate of outpatient surgery after holmium LASER enucleation of the prostate (HoLEP) for the treatment of BPH with and without the use of the MOSES 2.0 effect.

DETAILED DESCRIPTION:
HoLEP is in the process of becoming the new reference surgical treatment for BPH with the main advantages over monopolar transurethral resection (TURPm) and high approach adenomectomy (AVH): the significant reduction in morbidity perioperative period and therefore the reduction in the length of hospital stay. This reduction in length of stay has led to the development of outpatient care with encouraging results. The main cause of discharge failure on D0 is the persistence of postoperative hematuria requiring maintenance of bladder irrigation. MOSESTM 2.0 technology has the advantage of better hemostasis compared to the LASER LP100 currently used. The objective of this study is to evaluate the influence of MOSESTM 2.0 technology on the outpatient success rate in patients operated on for HoLEP for BPH.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 50 years old
* BPH whose symptoms require surgical management
* Preoperative prostate volume measured by ultrasound (suprapubic or transrectal) ≥ 40g
* IPSS score > 15 and Quality of Life score ≥ 3
* Maximum urinary output (Qmax) < 15 ml/sec

Exclusion Criteria:

* Inability to read or write French
* Patients with comorbidities contraindicating general anesthesia
* Patients not eligible for outpatient care according to French recommendations (high risk of complications after general anesthesia, place of residence more than 150 km from an emergency department, alone at home the night following the intervention) .
* History of BPH surgery
* History of prostate cancer
* Preoperative prostate volume measured by ultrasound (suprapubic or transrectal) < 40g
* Existence or history of urethral stricture
* Existence or suspicion of a "neurological" bladder
* Positive preoperative cytobacteriological examination not treated appropriately
* Adult patients subject to a legal protection measure or unable to express their consent
* Patients deprived of liberty by a judicial or administrative decision or hospitalized without consent or admitted to a health or social establishment for purposes other than research

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: * Patients who require HoLEP for Begnign Prostate Hypertrophy eligible for outpatient management
  * Patients having been managed by HoLEP (without MOSES 2.0) in ambulatory care since January 2016 in the urology department of the Bordeaux University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of patient who discharge on D0 (same day of his surgery) | baseline
Number of hour's hospitalization | baseline

SECONDARY OUTCOMES:
Number of hour's surgery time | baseline
Rate of enucleated prostate tissue By time treatment per patient | baseline
number of minutes use of the LASER during surgery | baseline
quantity of energy used during the intervention per patient | baseline
Intraoperative transfusion rate | baseline
Duration of post-operative sounding (hours) | baseline
Readmission rate within 48 hours of discharge from hospital | baseline
Mean change in IPSS before surgery and 3 months after surgery | 3 months after surgery
Mean change in QoL before surgery and 3 months after surgery | 3 months after surgery
Mean change in IIEF-5 before surgery and 3 months after surgery | 3 months after surgery
Mean change in ICIQ-short form score before surgery and 3 months after surgery | 3 months after surgery
Mean change in USP before surgery and 3 months after surgery | 3 months after surgery
Mean evolution of Qmax and post-void residual (RPM) before the intervention and at 3 months post-operative | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire ROBERT, PU-PH, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No